CLINICAL TRIAL: NCT05272098
Title: Comparative Effects of Myofascial Release Therapy and Endurance Training of Trunk Extensor Muscles on Pain, Disability and Muscle Endurance in Patients With Mechanical Back Pain.
Brief Title: Effects of Myofascial Release Therapy and Endurance Training on Mechanical Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/ 22/0101 Anum
Record Dates: First submitted 2022-02-20; First posted 2022-03-09 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Back Pain, Low
Keywords: Mechanical low back pain; myofascial release; endurance training; NPRS
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): myofascial release therapy
  Interventions: Other: Group A will receive myofascial release therapy + conventional physical therapy
- Group B (Active Comparator): endurance training of the trunk extensor muscles
  Interventions: Other: Group B will receive endurance training of the trunk extensor muscles + conventional physical therapy

INTERVENTIONS:
Other: Group A will receive myofascial release therapy + conventional physical therapy — myofascial release therapy (4 sessions per week). It soft, deep and non-manipulative form of treatment that involves the application of gentle pressure while stretching the body's connective tissue. A specialized form of touch, somatic sense, and specific body movement protocols are the three steps involved in the myofascial release therapy + hot pack (15min) + back care advice and postural modification. A total of 45 min session four times a week.
  Arms: Group A
Other: Group B will receive endurance training of the trunk extensor muscles + conventional physical therapy — It will be treated with endurance training of trunk extensor muscles. Erector spinae and latissimus dorsi will be included. The exercise protocol will be in four levels Bilateral shoulder left in prone position+ contralateral arm and leg lift in prone position+ both hands behind head and bilateral shoulder lift +bilateral shoulder lift with arm fully elevated + Hot pack (10 min) + back care advice and postural modification. A total of 45 min sessions four times a week.
  Arms: Group B

SUMMARY:
This study is a randomized clinical trial to determine the effects of myofascial release therapy versus endurance training of trunk extensor muscles on pain, disability and muscle endurance in patients with mechanical back pain. A sample of 24 patients will be taken and divided into two groups each with 12 patients. Group A will receive myofascial release therapy and conventional physical therapy while group B will endurance training of trunk extensors and the conventional physical therapy protocol. The conventional physical therapy protocol will include a hot pack, back care advice, and postural modifications. The session will be around 40 to 45 min for each patient with four sessions per week. A total of four-week treatment regime will be given to the patients and assessment of the patient's pain, disability, and endurance with NPRS (numeric pain rating scale), Rolland Morris Disability Questionnaire and Sorenson Test will be done at the baseline, after the completion of treatment at pre interventional and post interventional to observe the long-term effects. The data will be analyzed using SPSS.

DETAILED DESCRIPTION:
Mechanical low back pain is an injury of an anatomic structure in the low back. It accounts for 97% of cases arising from spinal structures such as bone ligaments, nerves, etc. In chronic low back pain, exercise therapy has become a first-line treatment and should be routinely used. Fascia is a form of connective tissue made up of collagen, surrounds the body parts, and resists tissue tensile load. Fascial injury and adhesions are common and can lead to pain, restricted motion, and swelling. The treatment of the fascial injury is necessary to relieve those symptoms. There are many treatments for mechanical back pain and this study focuses on two new treatment techniques for mechanical back pain. The first is the myofascial release therapy, a manual approach that focuses on the structural segmentation of fascia and involves the application of gentle pressure while stretching the body's connective tissues. The other treatment technique is the endurance training of the trunk extensor muscles that involve the treatment which is directed to endurance training of erector spinae and latissimus dorsi. The current study is novel in a way that there is limited literature about myofascial release therapy versus endurance training of trunk extensor muscles in patients with mechanical back pain. Both methods were employed to see if they improve pain along with accompanying disability and muscle endurance.

ELIGIBILITY:
Inclusion Criteria:

* History of mechanical low back pain
* Back pain without association with leg pain

Exclusion Criteria:

* Any bony, soft tissue or systemic disease

  * Pregnant females
  * Radiculopathy
  * Patient with spinal deformities and fractures

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
NPRS (numeric pain rating scale) | 4th week
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10) that best reflects the intensity of his/her pain 11-point numeric scale ranges from '0' representing no pain to 10 representing the worst imaginable pain.
Rolland Morris Disability Questionnaire | 4th Week
  It is designed to assess self-rated physical disability caused by low back pain. This scale has 24 points and each point will tell us about the disability of the patient pre and post-intervention. The score ranges from 0 (no disability) to 11, 18, or 24 (max. disability) depending on the questionnaire that is used.
Sorenson Test | 4th Week
  This test measures how many seconds the subject is able to keep the unsupported upper body (from the upper border of the iliac crest) horizontal, while placed prone with the buttocks and legs fixed to the couch by three wide canvas straps and the arms folded across the chest.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, Study Chair — Riphah International University; Anum Anwar, Principal Investigator — Riphah International University
Locations (1):
- Alkhaliq hospital Nishtar road, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ledford C. Spine Conditions: Mechanical and Inflammatory Low Back Pain. FP Essent. 2017 Oct;461:15-20. PMID 29019640
- [Background] Chien JJ, Bajwa ZH. What is mechanical back pain and how best to treat it? Curr Pain Headache Rep. 2008 Dec;12(6):406-11. doi: 10.1007/s11916-008-0069-3. PMID 18973732
- [Background] Urits I, Burshtein A, Sharma M, Testa L, Gold PA, Orhurhu V, Viswanath O, Jones MR, Sidransky MA, Spektor B, Kaye AD. Low Back Pain, a Comprehensive Review: Pathophysiology, Diagnosis, and Treatment. Curr Pain Headache Rep. 2019 Mar 11;23(3):23. doi: 10.1007/s11916-019-0757-1. PMID 30854609
- [Background] Hooten WM, Cohen SP. Evaluation and Treatment of Low Back Pain: A Clinically Focused Review for Primary Care Specialists. Mayo Clin Proc. 2015 Dec;90(12):1699-718. doi: 10.1016/j.mayocp.2015.10.009. PMID 26653300
- [Background] AAP Council on Communications and Media. Virtual Violence. Pediatrics. 2016;138(1):e20161298. Pediatrics. 2016 Oct;138(4):e20162399. doi: 10.1542/peds.2016-2399. No abstract available. PMID 27940893
- [Background] Rodriguez-Fuentes I, De Toro FJ, Rodriguez-Fuentes G, de Oliveira IM, Meijide-Failde R, Fuentes-Boquete IM. Myofascial Release Therapy in the Treatment of Occupational Mechanical Neck Pain: A Randomized Parallel Group Study. Am J Phys Med Rehabil. 2016 Jul;95(7):507-15. doi: 10.1097/PHM.0000000000000425. PMID 26745225
- [Background] Tantanatip A, Chang K-V. Myofascial Pain Syndrome. 2018.
- [Background] Sharan D, Rajkumar JS, Mohandoss M, Ranganathan R. Myofascial low back pain treatment. Curr Pain Headache Rep. 2014 Sep;18(9):449. doi: 10.1007/s11916-014-0449-9. PMID 25091133
- [Background] Jorgensen K. Human trunk extensor muscles physiology and ergonomics. Acta Physiol Scand Suppl. 1997;637:1-58. PMID 9246395
- [Background] Davis KG, Marras WS. The effects of motion on trunk biomechanics. Clin Biomech (Bristol). 2000 Dec;15(10):703-17. doi: 10.1016/s0268-0033(00)00035-8. PMID 11050352
- [Background] Salvetti Mde G, Pimenta CA, Braga PE, McGillion M. Prevalence of fatigue and associated factors in chronic low back pain patients. Rev Lat Am Enfermagem. 2013 Jan-Feb;21 Spec No:12-9. doi: 10.1590/s0104-11692013000700003. English, Portuguese. PMID 23459886